CLINICAL TRIAL: NCT02668419
Title: Neuromuscular Electrical Stimulation Improves Exercise Tolerance in Patients With Advanced Heart Failure on Continuous Dobutamine Use - A Randomized Controlled Trial
Brief Title: Electrical Stimulation Improves Exercise Tolerance in Patients With Advanced Heart Failure on Continuous Dobutamine Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Patricia Forstieri, PT, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13132413.0.0000.5505
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure; Ventricular Dysfunction, Left
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Patients in this group were subject to regular Physical Therapy Sessions in the hospital and each session consisted of breathing exercises and global active exercises of the upper and lower limbs in bed. The treatment was applied twice a day during the hospitalization period. The protocol was interrupted if the patient had signs or symptoms suggestive of poor tolerance to exercise.
  Interventions: Other: Physical Therapy Session
- Neuromuscular Electrical Stimulator (Experimental): Lower limb muscles of both legs were simultaneously stimulated using self adhesive surface rectangular electrodes. During all session period, the patients were maintained in the supine Fowler 45º position. The stimulation intensity was progressively increased according to the patient tolerance until a muscular contraction was observed. Stimulation was performed twice a day; the session duration was 60 min. Heart rate, blood pressure, respiratory rate and pulse oximetry were monitored throughout the sessions, in all patients.
  Interventions: Device: Neuromuscular Electrical Stimulator

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulator — Quadriceps and calf muscles of both legs were simultaneously stimulated using self adhesive surface rectangular electrodes. During all session period, the patients were maintained in the supine Fowler 45º position. Stimulation parameters were set up as follows: biphasic current of 40 Hz, 400-µs pulse duration, mode "on-time" 10s and "off-time" 20s and maximal amplitude of 60 mA. The stimulation intensity was progressively increased according to the patient tolerance until a muscular contraction was observed. Stimulation was performed twice a day; the session duration was 60 min.
  Other Names: NMES; Functional Electrical Stimulation (FES)
  Arms: Neuromuscular Electrical Stimulator
Other: Physical Therapy Session — each session consisted of breathing exercises and global active exercises of the upper and lower limbs in bed. The treatment was applied twice a day during the hospitalization period. The protocol was interrupted if the patient had signs or symptoms suggestive of poor tolerance to exercise: 1) cyanosis, pallor, dizziness, nausea or pre-syncope; 2) chest pain; 3) bradycardia; 4) a drop in systolic blood pressure >15 mmHg in comparison to baseline; 5) an excessive rise in systolic blood pressure defined as >200 mmHg; 6) a rise in diastolic blood pressure during exercise >110 mmHg; 7) fatigue rated ≥6/10 on the perceived exertion Borg scale (PEB); and/or 8) electrocardiographic signs of cardiac ischemia or ventricular arrhythmias.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine whether neuromuscular electrical stimulation can improve exercise tolerance for patients with heart failure and continuous dobutamine use in a hospital.

ELIGIBILITY:
Inclusion Criteria:

* Advanced heart failure (Stage D - Left ventricle ejection fraction <30%)
* New York Heart Association class III-IV
* Standard medical therapy for heart failure management
* Continuous inotropic infusion

Exclusion Criteria:

* Unstable angina pectoris
* Recent (6 months) acute coronary syndrome
* Arrythmias
* Chronic renal failure
* Diabetes Mellitus
* Peripheral vascular diseases
* Inability to walk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional capacity evaluated using the 6-minute walk test (6MWT) | Change from assessment at admission and at patient discharge
  Functional capacity was evaluated using the 6-minute walk test (6MWT), by a single evaluator blinded to the group allotment, in accordance with American Thoracic Society criteria.

SECONDARY OUTCOMES:
Change in the intravenous inotropic support dosage | Change from the first day of the protocol and patient discharge
  For all patients, the inotropic intravenous dose was adjusted daily by a single clinician (prescriber) blinded to the group allocation. Weaning from inotropic support was performed by the prescriber based on the improvement of clinical signs (level of consciousness, peripheral perfusion and blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Forestieri, PT, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No subject data will be made public. However, all participants were given the principal investigator's e-mail address and phone number in order to ask questions or receive their assessment results.